CLINICAL TRIAL: NCT02315560
Title: Foot Neuromodulation for Nocturnal Enuresis in Children
Brief Title: Foot Neuromodulation for Nocturnal Enuresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidi Stephany (Other)
Collaborators: Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction (Other)
Responsible Party: Sponsor-Investigator, Heidi Stephany, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO14080250
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Bedwetting
Keywords: bedwetting
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tibial Nerve Stimulation (Experimental): The subject/parents will be instructed to record a night-time voiding log specifying the number of incontinent episodes per night. This log is included in the Institutional Review Board application. Subjects/parents will fill out the log for a two week period prior to foot stimulation to determine a baseline average of nocturnal enuresis episodes, during the two week foot stimulation period to measure any acute effect on nocturnal enuresis episodes and finally during the two weeks after stimulation to evaluate any post-stimulation residual benefit
  Interventions: Device: TRANSCUTANEOUS ELECTRICAL NERVE STIMULATOR (TENS

INTERVENTIONS:
Device: TRANSCUTANEOUS ELECTRICAL NERVE STIMULATOR (TENS — electrical stimulation of the nerves in the foot on the incidence of nocturnal enuresis (bedwetting) in children

SUMMARY:
To determine the effects of electrical stimulation of the nerves in the foot on the incidence of nocturnal enuresis (bedwetting) in children

DETAILED DESCRIPTION:
Nocturnal Enuresis is a very common and difficult to treat problem in the pediatric population which can have significant negative impact on a child's quality of life. Apart from medications which can have significant side effects limiting their use, there is a lack of effective and safe treatment options for children with frequent nocturnal enuresis. If foot stimulation prior to bed does indeed improve the frequency of nocturnal enuresis, it may provide a safe and non-invasive therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 5 to 16 years old without any specific neurological disorder or urinary tract infection, clinically diagnosed as having nocturnal enuresis AT LEAST 4 episodes per month by history
2. Currently having no daytime overactive bladder symptoms, i.e. urinary frequency, urgency, or daytime incontinence
3. Having been assessed for and treated if applicable for behavioral etiologies of nocturnal enuresis - consuming excess fluids or specific bladder irritants
4. Having been assessed for and treated if applicable for constipation

Exclusion Criteria:

1. Children with known neurological disorders which may be contributing to nocturnal enuresis episodes
2. Children found through history to have significant behavioral causes of nocturnal enuresis including consumption of excessive fluids or known bladder irritants
3. Children with chronic constipation who are non-compliant with previous pharmacologic efforts to treat.
4. Children who are not adequately potty trained
5. Children with significant daytime symptoms of overactive bladder including frequency, urgency, and daytime incontinence

5. Children who do not tolerate initial stimulation training session in the urology clinic upon enrollment

6. Children with any implantable medical devices such as a pacemaker will be excluded from the study

Note: Any patient currently taking medication such as an anti-muscarinic or a tricyclic antidepressant for overactive bladder at time of enrollment will be eligible to participate and will be continued on their usual medication and dosage throughout the study.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Pittsburgh og UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tibial Nerve Stimulation
Started | 25
Completed | 22
Not Completed | 3
Not completed — noncompliance by subjects | 3

BASELINE CHARACTERISTICS:
Arm/Group | Tibial Nerve Stimulation
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 11.4 [7 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Nocturnal Enuresis
Description: To determine if foot stimulation can decrease nocturnal enuresis in children as measured by daily night-time voiding log. The outcome is the number of participants that had a clinical response with improvement of at least 1 wet night reduction during the 6-week stimulation period.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Foot Stimulation: The subject/parents will be instructed to record a night-time voiding log specifying the number of incontinent episodes per night. This log is included in the Institutional Review Board application. Subjects/parents will fill out the log for a two week period prior to foot stimulation to determine a baseline average of nocturnal enuresis episodes, during the two week foot stimulation period to measure any acute effect on nocturnal enuresis episodes and finally during the two weeks after stimulation to evaluate any post-stimulation residual benefit
  TRANSCUTANEOUS ELECTRICAL NERVE STIMULATOR (TENS: electrical stimulation of the nerves in the foot on the incidence of nocturnal enuresis (bedwetting) in children
Arm/Group | Foot Stimulation
Number analyzed (Participants) | 22
Participants | 16

2. Secondary Outcome: Quality of Life Questionnaire Scores
Description: The NLUTD/DES questionnaire (Neurogenic Lower Urinary Tract Dysfunction/Dysfunctional Elimination Syndrome) has been validated and is reliable for assessing lower urinary tract and bowel dysfunction. The questionnaire is scored using a 5-point Likert scale. The questionnaire consists of a total of 14 questions, each question asking about a symptom. Question #7 specifically addresses nocturnal enuresis. A score of 4 indicates severe symptoms, while a score of 0 indicates none. The maximum score is 52, indicating the most severe symptoms, while the minimum score of zero indicates zero symptoms. Scores of 11 or greater indicate bladder or bowel dysfunction.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Foot Stimulation
Number analyzed (Participants) | 22
units on a scale
  Pre-stimulation | 13.9 [5 to 35]
  Stimulation | 11.6 [5 to 33]
  Post-stimulation | 10.5 [2 to 28]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Foot Stimulation
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT02315560/Prot_SAP_000.pdf